CLINICAL TRIAL: NCT05084963
Title: A Phase 2a, Double-blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy, Safety, and Tolerability of IRL201104 in Adult Participants With Active Eosinophilic Esophagitis (EoE)
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of IRL201104 in Adults With Active Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revolo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVLO 121-04
Record Dates: First submitted 2021-09-30; First posted 2021-10-20 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — IRL201104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: IRL201104 Dose A (Experimental): IRL201104 IV on Days 0, 7, and 14
  Interventions: Drug: IRL201104
- Arm 2: IRL201104 Dose B (Experimental): IRL201104 IV on Days 0, 7, and 14
  Interventions: Drug: IRL201104
- Arm 3: Placebo (Placebo Comparator): Placebo IV on Days 0, 7, and 14
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IRL201104 — lyophilised powder for reconstitution for IV dosing
  Arms: Arm 1: IRL201104 Dose A; Arm 2: IRL201104 Dose B
Drug: Placebo — Matching placebo for IRL201104
  Arms: Arm 3: Placebo

SUMMARY:
The purpose of this study is to asses the efficacy, safety and tolerability of repeat doses of IRL201104 in Adult Participants with Active Eosinophilic Esophagitis (EoE)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old, inclusive, at the time of signing the informed consent form.
2. Documented diagnosis of EoE by endoscopy prior to screening. Note: Must include a demonstration of intraepithelial eosinophilic infiltration (peak cell count ≥ 15 eos/hpf [400×]) from esophageal biopsy specimens from endoscopy.
3. History (by participant report) of on average at least 2 episodes of dysphagia (with intake of solids off anti-inflammatory therapy) per week in the 4 weeks prior to screening, and on average at least 2 episodes of documented dysphagia per week during any 2 consecutive weeks (qualifying period) between screening and baseline; dysphagia is defined as trouble swallowing solid food, or having solid food stick, by participant report; and completed the DSQ on ≥ 70% of days during the qualifying period prior to baseline (Visit 1).
4. Must remain on a stabilized diet for at least 6 weeks prior to screening and during the course of the study; stable diet is defined as no initiation of single or multiple elimination diets or reintroduction of previously eliminated food groups.
5. Must be willing and able to continue any dietary therapy and/or medical regimens (including gastric acid suppression) in effect at the screening visit. There should be no change to these regimens during the study participation.
6. Willing and able to comply with all clinic visits and study-related procedures.
7. Able to understand and complete study-related questionnaires.
8. Provide signed informed consent.
9. Esophagogastroduodenoscopy (EGD) with photographs performed at screening (qualifying EGD), with a demonstration of intraepithelial eosinophilic infiltration (peak cell count ≥15 eos/hpf) in at least 2 of the 3 biopsied esophageal regions (proximal, mid, or distal).

Exclusion Criteria:

1. Prior participation in an IRL201104 clinical study.
2. Has any current disease of the gastrointestinal tract (aside from EoE) that may impact, in the investigator's opinion, the patient's EoE disease status. This includes, but not limited to: eosinophilic gastritis, eosinophilic enteritis, eosinophilic duodenitis, eosinophilic colitis, or proctitis; inflammatory bowel disease; or celiac disease.
3. Has other causes of esophageal eosinophilia or the following diseases: hypereosinophilic syndromes, Churg-Strauss vasculitis (eosinophilic granulomatosis with polyangiitis), or peripheral blood absolute eosinophil count of > 1500 eosinophils/μL.
4. Has presence of oral or esophageal mucosal infection of any type.
5. Has any condition affecting the esophageal mucosa or altering esophageal motility other than EoE.
6. History of achalasia, active Helicobacter pylori infection, Crohn's disease, ulcerative colitis, celiac disease, and prior esophageal surgery (with the exception of a surgical repair of an EoE complication).
7. Any esophageal stricture unable to be passed with a standard, diagnostic, adult (9 to 10 mm) upper endoscope or any critical esophageal stricture that requires dilation at screening; or dilation within 2 months prior to screening.
8. On a pure liquid diet or any mouth or dental condition that prevents normal eating.
9. Has initiated, discontinued, or changed dosage regimen of PPIs within the 4 weeks prior to the qualifying EGD, between the qualifying EGD and baseline visit (Visit 1), or anticipates changes in the use of PPI during the study. PPI must remain constant throughout the study.
10. History of bleeding disorders or esophageal varices.
11. Use of anticoagulants within 2 weeks prior to screening. Participants should not stop these agents solely to become eligible for entry into this study.
12. Treatment with an investigational drug within 2 months or within 5 half-lives (if known), whichever is longer, prior to screening.
13. Use of systemic corticosteroids within 3 months or swallowed topical corticosteroids within 6 weeks prior to screening.
14. Treatment with oral immunotherapy (OIT) within 6 months prior to screening.
15. Allergen immunotherapy (sublingual immunotherapy [SLIT] and/or subcutaneous immunotherapy [SCIT]), unless on a stable dose for at least 1 year prior to screening.
16. The following treatments within 3 months before the screening visit, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the study:

    Systemic immunosuppressive/immunomodulating drugs (eg, omalizumab, cyclosporine, mycophenolate-mofetil, interferon [IFN]γ, Janus kinase inhibitors, azathioprine, methotrexate, and other biologics that are ongoing [eg, dupilumab, benralizumab, mepolizumab, or vedolizumab]).
17. Diagnosed with active parasitic infection; or suspected parasitic infection, unless clinical and (if necessary) laboratory assessments have ruled out active infection before randomization.
18. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 1 month prior to screening.
19. Use of oral antibiotics/anti-infectives within 2 weeks prior to screening.
20. Known or suspected immunosuppression, including history of invasive opportunistic infections (eg, tuberculosis, non-tuberculous mycobacterial infections, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency, or prolonged infections suggesting an immunocompromised status, as judged by the investigator.
21. Known history of human immunodeficiency virus (HIV) infection.
22. Positive or indeterminate hepatitis B surface antigen (HBsAg) or hepatitis C antibody at screening.
23. Moderate or severe renal impairment (eGFR <60 mL/min/1.73 m2) or end stage renal disease.
24. Elevated transaminases (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) > 3 times the upper limit of normal (ULN) at screening.
25. History of malignancy within 5 years prior to screening, except completely treated in situ carcinoma of the cervix and completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin.
26. Any other medical or psychological condition including relevant laboratory abnormalities at screening that, in the opinion of the investigator, suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the participant as a result of his/her participation in this clinical study, may make the participant's participation unreliable, or may interfere with study assessments. The specific justification for participants excluded under this criterion will be noted in study documents (eg, chart notes, electronic case report form). These may include participant-reported alcohol or drug abuse and severe concomitant illness(es).
27. Planned or anticipated use of any prohibited medications and procedures (as described in the exclusion criteria) during study treatment.
28. Treatment with a live (attenuated) vaccine within 3 months prior to screening and/or treatment of a killed vaccine within 30 days prior to screening, until the end of the study with the exception of a coronavirus disease of 2019 (COVID-19) vaccine, as described in Section 9.2.1.
29. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
30. Women unwilling to use adequate birth control, if of reproductive potential* and sexually active. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 30 days after the last dose of study treatment. These include: hormonal contraceptives, intrauterine device, or double barrier contraception (ie, condom and diaphragm), or male partner with documented vasectomy.

    * For females, menopause is defined as at least 12 consecutive months without menses; to include laboratory confirmation of post-menopausal status (ie, a follicle stimulating hormone (FSH) of 2.25 U/mL must be documented). Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable; if documented, women with these conditions are not required to use additional contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weinreich, MD, PhD, Study Director — Senior Director, Revolo Biotherapeutics
Locations (22):
- United States (22):
  - Revolo Investigational Site, Little Rock, Arkansas
  - Revolo Investigational Site, Murrieta, California
  - Revolo Investigational Site, Centennial, Colorado
  - Revolo Investigational Site, New Port Richey, Florida
  - Revolo Investigational Site, Orlando, Florida
  - Revolo Investigational Site, Sandy Springs, Georgia
  - Revolo Investigational Site, Iowa City, Iowa
  - Revolo Investigational Site, Crowley, Louisiana
  - Revolo Investigational Site, Marrero, Louisiana
  - Revolo Investigational Site, Boston, Massachusetts
  - Revolo Investigational Site, Farmington Hills, Michigan
  - Revolo Investigational Site, Great Neck, New York
  - Revolo Investigational Site, Chapel Hill, North Carolina
  - Revolo Investigational Site, Durham, North Carolina
  - Revolo Investigational Site, Raleigh, North Carolina
  - Revolo Investigational Site, Mentor, Ohio
  - Revolo Investigational Site, Chattanooga, Tennessee
  - Revolo Investigational Site, Kingsport, Tennessee
  - Revolo Investigational Site, Baytown, Texas
  - Revolo Investigational Site, Harlingen, Texas
  - Revolo Investigational Site, Riverton, Utah
  - Revolo Investigational Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: IRL201104 4 mg; Arm 2: IRL201104 8 mg: IRL201104 IV on Days 0, 7, and 14
  IRL201104: lyophilised powder for reconstitution for IV dosing
Period: Overall Study
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Started | 12 | 12 | 12
Completed | 12 | 12 | 11
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) - includes all participants who were documented to have taken at least 1 dose of study treatment. Safety evaluations considered participants according to the actual treatment they received.
  (Note: One participant was randomised to Dose A but received Dose B for all 3 doses due to an error at the clinical site. The participant is considered under Dose A in the Full Analysis Set (FAS) as 'Randomized' and counted under Dose B in the SAS as 'Treated').
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo | Total
Number analyzed (Participants) | 11 | 13 | 12 | 36
Age, Continuous [Median (Full Range); unit: years] | 39 [21 to 57] | 42 [20 to 62] | 33 [20 to 52] | 38.5 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 6 | 10
  Male | 9 | 11 | 6 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 13 | 12 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Peak Esophageal Intraepithelial Eosinophil Count at Week 4 (Mean)
Description: The change from baseline in histologic eosinophil count in each treatment group will be summarized as the mean and Standard Deviation (SD)
Time Frame: 4 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: eosinophil count per high power field
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 12 | 12 | 12
eosinophil count per high power field | -9.2 (87.95) | -31.6 (68.09) | -7.8 (104.02)

2. Secondary Outcome: Absolute Change in Dysphagia Symptom Questionnaire (DSQ) Score From Baseline.
Description: The DSQ is used to measure the frequency and intensity of dysphagia. The DSQ scores can range from 0 to 84, with a lower score indicating less frequent or less severe dysphagia. The change from baseline in DSQ score in each treatment group will be summarized as the median, minimum, and maximum
Time Frame: 4 weeks
Population: Analysis performed on Full Analysis Set participants with non-missing DSQ data
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 10 | 12
score on a scale | -15.000 [-26.923 to 0.000] | -6.937 [-18.092 to 5.846] | -3.909 [-40.923 to 5.409]

3. Secondary Outcome: Percent of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of < 15 Eos/Hpf (Week 4)
Description: Percent of participants with a histologic eosinophil count of < 15 eos/hpf will be summarized for each treatment group
Time Frame: 4 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 1 | 1

4. Secondary Outcome: Percent Change in Peak Esophageal Intraepithelial Eosinophil Count (Eos/Hpf)
Description: The percent change from baseline in peak intraepithelial eosinophil count in each treatment group will be summarized as the mean and SD
Time Frame: 4 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 12 | 12 | 12
percent change | 31.061 (83.858) | -19.007 (39.716) | 44.306 (197.449)

5. Secondary Outcome: Treatment Emergent Adverse Events (TEAE)
Description: Number of participants who had a TEAE
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants | 6 | 7 | 7

6. Secondary Outcome: Safety Laboratory Data: Biochemistry
Description: Number of participants with treatment emergent clinically significant abnormal lab value.
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants
  Creatine Kinase | 1 | 0 | 0
  Alanine aminotransferase | 0 | 1 | 0
  Aspartate aminotransferase | 0 | 1 | 0
  Total Bilirubin | 0 | 1 | 0
  Indirect Bilirubin | 0 | 0 | 0
  Sodium | 0 | 0 | 0
  Total Protein | 0 | 0 | 0
  Potassium | 0 | 0 | 0
  Creatinine | 0 | 0 | 0
  Total Cholesterol | 0 | 0 | 0
  High-Density Lipoprotein | 0 | 0 | 0
  Low-Density Lipoprotein | 0 | 0 | 0
  Triglycerides | 0 | 0 | 0
  Glucose | 0 | 0 | 0
  Chloride | 0 | 0 | 0
  Blood Urea Nitrogen | 0 | 0 | 0
  Carbon dioxide | 0 | 0 | 0
  Calcium | 0 | 0 | 0
  Alkaline phosphatase | 0 | 0 | 0
  Uric acid | 0 | 0 | 0
  Albumin | 0 | 0 | 0
  Lactate dehydrogenase | 0 | 0 | 0

7. Secondary Outcome: Safety Laboratory Data: Coagulation
Description: Number of participants with treatment emergent clinically significant abnormal lab value
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants
  Activated partial thromboplastin time | 0 | 1 | 0
  Prothrombin time | 0 | 1 | 0

8. Secondary Outcome: Safety Laboratory Data: Hematology Panel
Description: Number of participants with treatment emergent clinically significant abnormal value [Hemoglobin, Hematocrit, red blood cells count, white blood cell count, red cell indices, platelet count and white blood cell differential (neutrophil, lymphocyte, monocyte, eosinophil, and basophil)].
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants | 0 | 0 | 0

9. Secondary Outcome: Safety Laboratory Data: Urinalysis Panel
Description: Number of participants with treatment emergent clinically significant abnormal value (Color, Glucose, Red blood cells, Clarity, Blood, Hyaline and other casts, pH, Bilirubin, Bacteria, Specific gravity, Leukocyte esterase, Epithelial cells, Ketones, Nitrite, Crystals, Protein, White blood cells, Yeast).
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants | 0 | 0 | 0

10. Secondary Outcome: 12-Lead ECG
Description: Number of participants with treatment emergent clinically significant abnormal value (Ventricular Rate, PR Interval, RR Interval, QRS Duration, QT Interval, QTcF Interval).
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants | 0 | 0 | 0

11. Secondary Outcome: Physical Exam
Description: Number of participants with treatment emergent clinically significant abnormal value [Body Systems: head, eyes, ears, nose and throat (HEENT); cardiovascular, respiratory, gastrointestinal, dermatological, musculoskeletal, nervous systems, lymph nodes and general appearance].
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants | 0 | 0 | 0

12. Secondary Outcome: Vital Signs
Description: Number of participants with treatment emergent clinically significant abnormal value (systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature).
Time Frame: 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
Number analyzed (Participants) | 11 | 13 | 12
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to week 8
Description: Safety Analysis Set - includes all participants who were documented to have taken at least 1 dose of study treatment. Safety evaluations will consider participants according to the actual treatment they received.
Arm/Group | Arm 1: IRL201104 4 mg | Arm 2: IRL201104 8 mg | Arm 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 6/11 | 7/13 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: IRL201104 4 mg (N=11) | Arm 2: IRL201104 8 mg (N=13) | Arm 3: Placebo (N=12)
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine phosphatase increased (Investigations) | 1 | 0 | 0
Type IIb hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05084963/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT05084963/SAP_001.pdf